CLINICAL TRIAL: NCT02975778
Title: Prediction of Pain During Old People Care Measured by Skin Conductance
Acronym: DOLOAGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Budgetary and operational issues
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2016/27; 2016-A00709-42 (Other: ANSM)
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Pain
Keywords: 65 years old
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aged, 65 and over (Experimental)
  Interventions: Device: Pain Monitor™

INTERVENTIONS:
Device: Pain Monitor™ — Pain measured by Pain Monitor™

SUMMARY:
The purpose of the project is to validate the use of Pain Monitor™ device, not invasive and simple of employment, for old people able to answer to a digital scale of pain intensity.

The main objective is to develop and to validate a model of prediction of the pain in old subject at the time of the care, using the measure of variation of the skin conductance.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized patient;
* patient over 65 years of age;
* communicating, without cognitive impairment;
* having to undergo an act presumed to be painful during which the patient's mobility is limited: nursing care (removal of a drain, dressing of a chronic wound, urinary catheterization, etc.), medical examination, etc.;
* benefiting from a social security scheme or having rights;
* having given their prior informed written consent;
* person able to read.

Exclusion Criteria:

* cutaneous anomaly on the site of measure;
* pacemaker or internal defibrillator;
* extremities twitching;
* Treated by neostigmine.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

PRIMARY OUTCOMES:
Correlation between Number of pics of skin conductance per second measured by Pain Monitor™ device with Numerical visual scale score for pain | 14 days

SECONDARY OUTCOMES:
Hospital Anxiety and Depression (HAD) score | 14 days
Percentage of efficient poses of Pain Monitor | 14 days
Percentage of patient refusal to use of the Pain monitor | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fischler, MD, PhD, Study Director — Hopital Foch
Locations (2):
- France (2):
  - Maison Médicale Jeanne Garnier, Paris
  - Hopital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No